CLINICAL TRIAL: NCT07109401
Title: Perioperative Tislelizumab for Resectable Small Cell Lung Cancer in Stage IIB-IIIB: A Phase 2 Trial
Brief Title: Perioperative Immunotherapy for Resectable Limited-Stage SCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Director in the Department of Thoracic Surgery, FUSCC, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECTOP-1033
Record Dates: First submitted 2025-07-24; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Perioperative Immunotherapy; Limited Stage Lung Small Cell Carcinoma; Resectable Small Cell Lung Cancer
MeSH Terms: interventions — tislelizumab; Cisplatin; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perioperative Tislelizumab combined with Etoposide and Platinum-based Chemotherapy (Experimental): Neoadjuvant therapy: Tislelizumab 200mg, i.v., q3w, 2-4 cycles; Cisplatin 75mg/m2, d1 or Carboplatin AUC5-6, d1 + Etoposide 100mg/m2, d1-3, q3w, 2-4 cycles.
  Those resectable after neoadjuvant therapy will be treated with radical surgery.
  Adjuvant therapy: Patients received radical surgery will be treated with Tislelizumab plus platinum-etoposide therapy (the total cycle of perioperative chemotherapy is four), followed by Tislelizumab monotherapy for one year.
  Interventions: Drug: Tislelizumab (BGB-A317) Plus Chemotherapy (Cisplatin/Carboplatin and Etoposide)

INTERVENTIONS:
Drug: Tislelizumab (BGB-A317) Plus Chemotherapy (Cisplatin/Carboplatin and Etoposide) — Neoadjuvant therapy: Tislelizumab + Cisplatin or Carboplatin + Etoposide; Adjuvant therapy: Tislelizumab + Cisplatin or Carboplatin + Etoposide (the total cycle of perioperative chemotherapy is four), followed by Tislelizumab monotherapy for one year.

SUMMARY:
For limited-stage small cell lung cancer (SCLC), surgical treatment is recommended for patients with T1-2N0M0 (I-IIA) by guidelines. However, whether perioperative immunotherapy extends radical surgery to stage IIB-IIIB patients with improved survival remains elusive.

This is a phase II, single-arm study to evaluate the efficacy and safety of neoadjuvant Tislelizumab + chemotherapy (Cisplatin/Carboplatin + Etoposide) followed by radical surgery and adjuvant Tislelizumab ± chemotherapy for patients with limited-stage SCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent and understand and agree to comply with the study requirements and assessment schedule;
2. Aged 18-75 years at the time of signing the informed consent form;
3. Pathologically (histologically or cytologically) confirmed diagnosis of small cell lung cancer;
4. Limited-stage disease (stage IIB-IIIB according to AJCC 8th edition) assessed by bronchoscopy, PET-CT, endobronchial ultrasound (EBUS), mediastinoscopy, or percutaneous biopsy, deemed resectable with curative intent (R0 resection) by the investigator.

   TNM staging includes T3-4 (N0 only) or N1-2 (any T) and M0, where T4 is limited to tumors >7 cm in diameter; Patients with tumors invading the diaphragm, mediastinum, heart, great vessels, trachea, recurrent laryngeal nerve, esophagus, vertebral body, carina or having separate tumor nodules in different ipsilateral lobes are excluded. N2 is limited to single station and non-bulky.
5. No prior radiotherapy, chemotherapy, immunotherapy, surgery or other systemic treatments;
6. ECOG PS score of 0-1;
7. Expected survival must be >3 months;
8. Adequate bone marrow reserve and organ function within 30 days prior to enrollment meeting criteria for receiving platinum-based doublet chemotherapy;
9. No contraindications for immunotherapy.

Exclusion Criteria:

1. Tumor histopathology indicates non-small cell lung cancer (NSCLC);
2. Presence of clinically inactive or active brain metastases;
3. Any history of interstitial lung disease (ILD) (including pulmonary fibrosis or radiation pneumonitis), current ILD, or suspicion of such diseases based on imaging during screening;
4. Receiving systemic corticosteroid therapy within 14 days prior to the first dose of study drug;
5. Previous radiotherapy, chemotherapy, immunotherapy, surgery, or other systemic treatments;
6. Any active malignancy within 2 years prior to enrollment;
7. Women who are pregnant, breastfeeding, or planning to become pregnant during the study period;
8. Uncontrolled or significant cardiovascular disease at the time of enrollment;
9. Active or previously recorded autoimmune or inflammatory diseases before enrollment;
10. History of active primary immunodeficiency disorders;
11. Presence of active infections;
12. Active bleeding disorders within ≤6 months prior to administration of the study drug, including gastrointestinal bleeding evidenced by hematemesis, severe hemoptysis, or melena;
13. Non-healing wounds, active peptic ulcers, or fractures;
14. Any condition that the investigator deems makes the patient unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
One-year Event-free Survival Rate (1-year EFS Rate) | Up to 12 months
  The proportion of patients who have not experienced an EFS event within 1 year after the first administration of the study drug. EFS (Event-Free Survival) is defined as the time from the first dose of study treatment until the first occurrence of any of the following events: objectively documented disease progression and inability to undergo radical surgery, local recurrence, distant metastasis, or death from any cause (whichever occurs first). EFS is assessed by investigators based on RECIST v1.1 (Response evaluation criteria in solid tumors v1.1) criteria within the radical curative therapy analysis set.

SECONDARY OUTCOMES:
Event-free Survival (EFS) | up to 60 months
  Event-Free Survival (EFS) - defined as the time from the first dose of study treatment until the first occurrence of any of the following events: objectively documented disease progression and inability to undergo radical surgery, local recurrence, distant metastasis, or death from any cause (whichever occurs first).
Overall Survival (OS) | up to 60 months
  Overall Survival - defined as the time from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.
Objective Response Rate (ORR) | Up to 12 months
  Objective Response Rate (ORR) - defined as the proportion of patients who achieve a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR), as assessed by investigators according to RECIST v1.1 criteria.
Disease Control Rate (DCR) | Up to 12 months
  Disease Control Rate (DCR) - defined as the proportion of patients who achieve a Best Overall Response (BOR) of Complete Response (CR), Partial Response (PR), or Stable Disease (SD), as assessed by investigators according to RECIST v1.1 criteria.
Pathological Complete Response (pCR) Rate | Up to 12 months
  Pathological Complete Response (pCR) Rate - defined as the proportion of patients who have no residual tumor in the resected primary tumor site and all resected lymph nodes after neoadjuvant therapy among those who underwent surgical resection.
Major Pathological Response (MPR) Rate | Up to 12 months
  Major Pathological Response (MPR) Rate - defined as the proportion of patients who have ≤10% residual viable tumor cells in the resected primary tumor site and all resected lymph nodes after neoadjuvant therapy among those who underwent surgical resection.
Pathological Downstaging Rate | Up to 12 months
  Pathological Downstaging Rate - defined as the proportion of patients who undergo surgical resection after neoadjuvant therapy and have a postoperative pathological stage that is lower than their baseline clinical tumor stage and/or lymph node involvement.
R0 Resection Rate | Up to 12 months
  R0 Resection Rate - defined as the proportion of patients who achieve complete tumor resection (negative margins with no residual tumor cells) among those who underwent surgical resection after neoadjuvant therapy.
Clinical Downstaging Rate | Up to 12 months
  Clinical Downstaging Rate - defined as the proportion of patients who have a reduction in tumor size and/or lymph node involvement in their clinical tumor stage after neoadjuvant therapy compared to their baseline clinical tumor stage before surgery.
Surgical Resection Rate | Up to 12 months
  Surgical Resection Rate - defined as the proportion of patients who undergo surgical resection after neoadjuvant therapy.
Incidence of Treatment-emergent Adverse Event (TEAE) and Immune-related Adverse Event (IrAE) | Up to 60 months
  The incidence of TEAE and IrAE will be assessed by monitoring adverse events (AEs) and serious adverse events (SAEs) as described in the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0, and by incorporating relevant physical examinations, electrocardiograms (ECGs), and laboratory tests as needed.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
The clinical data including patient characteristics, CT images and pathology images.